CLINICAL TRIAL: NCT03684213
Title: The Effect of Local Antioxidant Therapy on Racial Differences in Vasoconstriction
Brief Title: Local Antioxidant Therapy Vasoconstriction Effects in Different Races
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Matthew Brothers, Associate Professor / Associate Chair for Graduate Programs in Exercise Science and Kinesiology Director of the Integrative Vascular Physiology Laboratory, The University of Texas at Arlington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-0647
Record Dates: First submitted 2018-09-17; First posted 2018-09-25 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; Vasoconstriction
Keywords: Racial Differences; Oxidative Stress; Antioxidant; Microvasculature
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Norepinephrine; Ascorbic Acid; NG-Nitroarginine Methyl Ester

STUDY DESIGN:
Intervention Model Description: Each subject has one control site and three experimental sites concurrently tested within the same study using intradermal microdialysis on the dorsal forearm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Control (Norepinephrine) (Active Comparator): Subjects will be administered norepinephrine at varying concentrations (10^-2 to 10^-8 M phenylephrine) at a rate of 2 microliters/minute for 10 minutes at each dose to construct a dose-response curve.
  Interventions: Drug: Control (Norepinephrine)
- Norepinephrine + Ascorbic Acid (Experimental): Subjects will be coinfused with the same norepinephrine concentrations as the control arm and ascorbic acid (Vitamin C; 10 mM) at the same rate and for the same time as the control arm.
  Interventions: Drug: Norepinephrine + Ascorbic Acid
- Norepinephrine + L-NAME (Experimental): Subjects will be coinfused with the same norepinephrine concentrations as the control arm and L-NAME (Nω-Nitro-L-arginine methyl ester hydrochloride; 20 mM) at the same rate and for the same time as the control arm.
  Interventions: Drug: Norepinephrine + L-NAME
- Norepinephrine + L-NAME + Ascorbic Acid (Experimental): Subjects will be coinfused with the same norepinephrine concentrations as the control arm and combined L-NAME (Nω-Nitro-L-arginine methyl ester hydrochloride; 20 mM) and ascorbic acid (Vitamin C; 10 mM) at the same rate and for the same time as the control arm.
  Interventions: Drug: Norepinephrine + L-NAME + Ascorbic Acid

INTERVENTIONS:
Drug: Control (Norepinephrine) — This intervention is aimed at assessing the vascular responsiveness to norepinephrine, an alpha 1-agonist, in white and black men and women across a series of ascending dose concentrations.
  Arms: Control (Norepinephrine)
Drug: Norepinephrine + Ascorbic Acid — This intervention is meant to globally assess the impact of oxidative stress on vasoconstrictor responses by scavenging numerous oxidative molecules.
  Arms: Norepinephrine + Ascorbic Acid
Drug: Norepinephrine + L-NAME — This intervention is meant to assess the impact of endothelium-derived nitric oxide on vasoconstrictor responses by inhibiting production of this source of nitric oxide.
  Arms: Norepinephrine + L-NAME
Drug: Norepinephrine + L-NAME + Ascorbic Acid — This intervention is meant to assess the combined impact of scavenging oxidative stress and inhibiting endothelium-derived nitric oxide on vasoconstrictor responses.
  Arms: Norepinephrine + L-NAME + Ascorbic Acid

SUMMARY:
Cardiovascular disease (CVD) afflicts nearly one-third of the adult population with all races and ethnicities represented in CVD prevalence. Unfortunately, a disparity exists such that the black population (BL) is disproportionately affected compared to other groups, including the white population (WH). While the underlying cause of this disparity is multifactorial, vascular dysfunction (i.e., impaired vasodilation and/or augmented vasoconstriction) is a key contributor. As has been previously observed, BL exhibit a heightened vasoconstrictor response to both pharmacological (e.g., alpha-adrenergic receptor agonists) and environmental (e.g., cold pressor test) stimuli compared to their WH counterparts. Additionally, reactive oxygen species (ROS) and the subsequent reduction in nitric oxide (NO) bioavailability may partially mediate this response. Our laboratory has recently observed (UTA IRB 2016-0268) that the small blood vessels in the skin (cutaneous microvasculature) in BL, but otherwise healthy individuals, produce an impaired blood flow response to local heating when compared to age-, body mass index (BMI)-, and gender-matched WH. However, pre-treatment of the cutaneous microvasculature with various antioxidants abolishes this skin blood flow difference. These antioxidant drugs inhibit possible sources of ROS, which, as mentioned, maybe mediating the heightened vasoconstrictor response in BL. However, this has not been investigated in this population and thus remains unknown. Therefore, the purpose of this study proposal is to test the following hypotheses: 1) BL will have a greater reduction in cutaneous blood flow in response to local administration of Norepinephrine (alpha1-adrenergic and alpha 2-adrenergic receptor agonist) relative to WH. 2) This greater reduction in the BL population will be related to elevated oxidative stress and subsequent reduction in bioavailability of the potent vasodilator Nitric oxide.

DETAILED DESCRIPTION:
Collectively, these studies will provide novel data and insight into the impact of heightened vasoconstrictor responses in BL on vascular function. Interested participants will be asked to come in the fasted state (a minimum of 3 hr since the last meal) and to have refrained from alcohol, caffeine, and physical activity for 24 hr. We will first review the inclusion/exclusion criteria and discuss the informed consent form including an oral explanation of the study purpose, experimental procedures and measurements, and potential risks and benefits associated with participation. Prior to any screening/testing, all subjects will provide written, informed consent. A medical health history questionnaire will then be completed by the subject and subsequently reviewed by the research team to determine eligibility. For the qualified participants, to test the aforementioned hypotheses, we will use laser Doppler to assess the skin blood flow response to local administration of the sympathomimetic drug-norepinephrine which is an alpha-1 and alpha-2 -adrenergic receptor agonist. Each participant will be instrumented with four cutaneous microdialysis fibers in the skin of the non-dominant forearm. Each of the following conditions will be randomly assigned to an individual microdialysis site. Experimental sites will then be infused with their respective vasoactive agents at a rate of 2 μl/min for a 30 min wash-in period. Site 1: This site will serve as the control site and will receive lactated Ringer's (saline solution). Site2: This site will receive 20 mM L-NAME (Nω-Nitro-L-arginine methyl ester hydrochloride, Sigma Aldrich) to inhibit nitric oxide production by nitric oxide synthase. This site will then be infused with no more than 10mM of norepinephrine to elicit vasoconstriction. Site 3: This site will receive 10 mM Ascorbic Acid which serves as a non-selective antioxidant. Ascorbic acid is commonly known as Vitamin C. This site will then be infused with no more than 10mM of norepinephrine to elicit vasoconstriction. Site 4: This site will receive a combination of 20mM L-NAME + 10 mM ascorbic acid. This site will then be infused with incremental doses of 10-8M - 10-2M of norepinephrine to elicit vasoconstriction. This dose and approach is commonly utilized in these types of studies. After the 30-min wash-in period, 15-min of baseline data will be collected with local heaters set to 33°C(91.4°F). After 15 min of baseline data collection, the perfusate at each site will be switched to various concentrations of norepinephrine combined with the respective vasoactive agent for each site-incremental doses of 10-8M - 10-2M (no more than 10mM(10-2M) at a rate of 2 μl/min for a brief period (no more than 6-min each dose) to quantify the level of vasoconstriction at each site. The order of the procedure will be as follows: 1. Instrumentation with membranes. 2. Wash-in perfusion with vasoactive agent at respective site (each site will receive its respective vasoactive agent simultaneously). Temperature set at 33°C(91.4°F). 3. Baseline data collection. Temperature set at 33 degree C(91.4°F). 4. Switch to Norepinephrine + combined vasoactive agent (for each respective site) infusion. Temperature set at 33 degree C(91.4°F). 5. Repeat step 4 for each concentration of norepinephrine used. As commonly done in these types of studies there will not be any flushes of Ringer's solution between doses of NE. In addition we will also measure blood flow in the brachial artery using Doppler ultrasound during resting conditions as well as during a standard flow mediated dilation (FMD) protocol. This includes inflating a blood pressure cuff to suprasystolic pressures (pressure slightly above the participant's systolic blood pressure) for 5 min and making continuous blood flow measures before and after release of the cuff. This will be performed on the upper arm in the brachial artery. This is a standard procedure used in numerous clinical investigations to estimate endothelial function with no reports of injury or adverse events. Subject Participation: During the course of the study, a subject may decide not to participate in a particular experimental measurement or procedure and therefore, this portion of the protocol will not be completed. However, all other measurements and procedures will be performed. This will not affect the scientific value of the subject's participation as each experimental measurement and procedure provides important and in most cases independent information.

ELIGIBILITY:
Inclusion Criteria:

* Individuals (ages 18-35, both genders) will be recruited from the greater Arlington area to participate in the study.
* Must self-report both parents as either African American or Caucasian American.

Exclusion Criteria:

* Individuals who have donated more than 550 ml of blood within the past 8 weeks will not have blood drawn from them in this protocol. However, if they remain interested in the study, and otherwise meet the inclusion criteria, than we may still opt to proceed with data collection.
* Individuals with cardiovascular, neurological, and/or metabolic illnesses will be excluded from participating as well as individuals with a history of various diseases of the microvasculature including Reynaud's disease, cold-induced urticaria, cryoglobulinemia, etc.
* Subjects currently taking any prescription medications and individuals with a body mass index about 30 kg/m2) will be excluded.
* Pregnant subjects and children (i.e. younger than 18) will not be recruited for the study. Eligible females will be scheduled for days 2-7 of their menstrual cycle to account for hormonal effects on blood flow. A regular menstrual cycle is required to identify and schedule the study for the low hormone period, therefore females who lack a regular cycle will be excluded from the study. Females currently taking birth control are eligible, as long as they can be scheduled during a low-hormone "placebo" week. If their hormone do not contain a placebo week than these individuals will not be eligible for data collection. Females who are breast-feeding will also be eligible as there are no systemic or lasting effects of the proposed vasoactive agents.
* Given that smoking can affect the peripheral vasculature, current smokers and individuals who regularly smoked (>1 pack per two weeks) within the prior 2 years will be excluded

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-08 (Actual)

PRIMARY OUTCOMES:
Vasoconstrictor Responsiveness to Norepinephrine using Laser Doppler Fluxmetry | Through study completion, an average of 1 Year
  Establish heightened vasoconstriction to norepinephrine stimulation in black men and women with a focus on black women. Following the local infusion of norepinephrine, the changes in blood flux will be quantified using laser Doppler fluxmetry. All changes in flux will be normalized and reported as a percentage of baseline flux.
Role of Oxidative Stress in Heightened Vasoconstriction using Laser Doppler Fluxmetry | Through study completion, an average of 1 Year
  Determine to what degree global oxidative stress and differences in endothelial nitric oxide play a role in heightened vasoconstriction. Following the local infusion of norepinephrine combined with either Ascorbic Acid, L-NAME, or L-NAME with Ascorbic Acid, the changes in blood flux will be quantified using laser Doppler fluxmetry. All changes in flux will be normalized and reported as a percentage of baseline flux.

CONTACTS AND LOCATIONS:
Locations (1):
- Science and Engineering Research and Innovation Building, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No